CLINICAL TRIAL: NCT06892275
Title: The FYI on MRI: A Multilevel Decision Support Intervention for Screening Breast MRI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: STUDY00008530
Record Dates: First submitted 2025-03-11; First posted 2025-03-24 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Breast Neoplasm Female; Early Detection of Cancer; Hereditary Breast and Ovarian Cancer Syndrome; Magnetic Resonance Imaging
MeSH Terms: conditions — Hereditary Breast and Ovarian Cancer Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Enhanced Usual Care (Active Comparator): Participants in this arm will be mailed a letter with their estimated lifetime risk for breast cancer per the NCI Breast Cancer Risk Assessment Tool (BCRAT), information about screening breast MRI, and instructions for contacting the nurse practitioner (NP) at the Ralph Lauren Center (RLC) with questions.
  Interventions: Behavioral: Enhanced Usual Care
- Decision Support (Experimental): Participants in this arm will receive the same letter as those in the Enhanced Usual Care arm. In addition, they will be sent the decision aid via mail or email (as preferred).
  Interventions: Behavioral: Enhanced Usual Care; Behavioral: Decision Support

INTERVENTIONS:
Behavioral: Enhanced Usual Care — Risk assessment and notification, referral to nurse practitioner (NP) at the Ralph Lauren Center (RLC)
Behavioral: Decision Support — The decision aid describes two different breast cancer screening plans: (1) annual mammography only; and (2) annual mammography plus annual breast MRI. The decision aid provides balanced information about breast MRI, including its risks, limitations, and benefits.
  Arms: Decision Support

SUMMARY:
The purpose of this study is to test the impact of a multilevel decision support intervention on informed decisions about breast MRI among high-risk Black and Latina women. Participants (N=80) will be randomized to (1) enhanced usual care (risk assessment + referral to nurse practitioner) or (2) decision support (enhanced usual care + decision aid). Assessments will take place at baseline (T0) and 1-month post-intervention (T1). The primary outcome is informed decisions about breast MRI at T1.

DETAILED DESCRIPTION:
The aim of this study is to evaluate whether the decision support intervention produces a clinically significant change in informed decisions about breast MRI. An informed decision is defined as a decision that is made with sufficient knowledge, and is in line with the person's preferences. The investigators will achieve this aim through a randomized controlled trial. This trial adheres to well-established design and reporting criteria for behavioral intervention studies to ensure patient safety and examine trial outcomes.<br> <br> Research Design. The main hypothesis is that participants receiving the decision support intervention will be more likely to make an informed decision about breast MRI v. participants receiving enhanced usual care. To test this hypothesis, participants (N=80) will be randomized to one of two arms: (1) enhanced usual care (breast cancer risk assessment + referral to nurse practitioner) or (2) decision support (enhanced usual care + decision aid). This design will allow us to examine the effect of decision support above and beyond breast cancer risk assessment and notification.<br> <br> Participants and Eligibility. The investigators will enroll a total of 80 Black and Latina women with high risk for breast cancer, defined as ≥20% lifetime risk for breast cancer. Participants will be recruited from the Ralph Lauren Center (RLC), a community-based clinic in Washington, DC, affiliated with the Georgetown Lombardi Comprehensive Cancer Center. <br> <br> Access. Participants must adequately speak English or Spanish to participate; the investigators will include those who are bilingual. To support access for women who report Spanish as their primary language, a bilingual/bicultural research assistant will approach, recruit, and complete assessments with these participants and provide additional study support as needed. In addition, all study materials will be available in both English and Spanish.<br> <br> Recruitment and Enrollment. During intake interviews for new RLC patients, navigators will administer the NCI Breast Cancer Risk Assessment Tool (BCRAT) via phone, enter responses into the BCRAT website in real-time, calculate lifetime breast cancer risk, and document BCRAT results in RLC's HIPAA-compliant, web-based patient tracking platform (RIPPLE©). The investigators estimate that this process will take <5 minutes to complete. The BCRAT provides estimated lifetime risk for breast cancer to inform use of breast MRI, and will be used to determine study eligibility. At this point, all women will continue routine mammography navigation. Women will receive mammogram results via mail; study staff will confirm normal mammogram results via the EMR. A research assistant (RA) will then contact high-risk women with a negative mammogram via phone, confirm eligibility, introduce the study, answer any questions, obtain verbal informed consent, and conduct the baseline assessment. Participants will be randomized immediately following the baseline assessment.<br> <br> Intervention Conditions. Participants in the Enhanced Usual Care arm will be mailed a letter with their estimated lifetime risk for breast cancer per the NCI Breast Cancer Risk Assessment Tool (BCRAT), information about screening breast MRI, and instructions for contacting the nurse practitioner (NP) at RLC with questions. Participants in the Decision Support arm will receive the same letter as those in the Enhanced Usual Care arm. In addition, they will be sent a decision aid via mail or email (as preferred). The decision aid describes two different breast cancer screening plans: (1) annual mammography only; and (2) annual mammography plus annual breast MRI. The decision aid provides balanced information about breast MRI, including its risks, limitations, and benefits. The decision aid will emphasize that there is no 'correct' decision and women should pick the plan that is right for them. It will also include: (1) facts about breast cancer and breast cancer risk (e.g., what does it mean to be at high risk, factors contributing to breast cancer risk, etc.); (2) answers to frequently asked questions about breast cancer screening; (3) an interactive exercise to clarify screening preferences; (4) information about cost/insurance coverage for breast cancer screening; and (5) instructions for accessing breast cancer screening (both mammogram and MRI) via RLC. The decision aid will emphasize that the nurse practitioner (NP) at RLC can provide a referral for mammogram and/or MRI to interested patients.<br> <br> Randomization. A computer-generated randomization table will be used to assign participants (N=80) to intervention conditions (n=40 per condition). Randomization will be stratified by race/ethnicity in random block sizes of 4, 8, or 12 to ensure balance across conditions.<br> <br> Measures. System-level data (i.e., CBCC patients navigated, high-risk women identified) will be obtained via EMR review. Patient-level data will be obtained via EMR review and participant self-report. Participants will complete self-report measures at baseline (T0) and 1-month post-intervention (T1) in-person or via phone with the assistance of a bilingual/bicultural RA (as preferred). The timing of the T1 assessment was selected in order to provide enough time for the intervention participants to receive/use the decision aid. Thus, the T1 survey allows for examination of the short-term effects of the decision aid. All measures will be available in English and Spanish. As noted above, a certified translator will be used to create a Spanish-language version.<br> <br> Hypotheses. The investigators will test the following two hypotheses:<br>

1. H1: Intervention (v. enhanced usual care) participants will be more likely to make an informed decision about breast MRI.<br>
2. H2: Intervention (v. enhanced usual care) participants will have greater decision satisfaction and less decisional conflict.<br> <br> Clinical trial management. This trial uses timed delivery of assessments. The investigators use a clinical trial data management system at the Georgetown Lombardi Comprehensive Cancer Center (GLCCC) Data Management Core (DMC) to facilitate and monitor trial operational flow and processes. At randomization, the DMC prepares a transition packet with background information about each participant's age, race/ethnicity, and risk for breast cancer. It is transmitted to the investigators, who ensure that all participants are mailed the appropriate materials for their randomization condition. A research assistant (RA) will document the distribution of all study materials and any contact by participants (i.e., with questions, to withdraw from the study, etc.). RLC's NP will also report to the study team if she completes any appointments with study participants. These data will be remotely uploaded into the DMC system and reviewed by the investigators for quality control, protocol monitoring, and fidelity.<br> <br> Distress monitoring protocol. The RA and navigator may experience some challenges addressing participants' emotional distress, unresponsiveness, and other problems. Participants may also have needs for resources beyond decision support. As recommended, the investigators have a well-established back-up protocol in place. In training, the RA and navigator will receive instruction and a referral card with the name, 24/7 telephone number, and e-mail of the PI (a licensed clinical psychologist) with instructions to contact her in the event of a crisis or emergency. The PI will provide consultation, emotional and logistic support, and referral for clinical services as needed.<br> <br> Retention. The investigators will deliver telephone and e-mail reminders and use flexible scheduling to promote retention. The investigators will also make multiple attempts to reach participants for intervention and data collection. After reaching an IRB-defined threshold, the investigators will mail a letter encouraging participants to contact us to complete the trial.<br> <br> Expected Outcomes. Upon completion of this RCT, the investigators will have data on the impact of the multilevel decision support intervention on informed decisions about breast MRI. Regardless of the effect of the decision aid on the outcomes of interest, the enhanced usual care arm will be a viable intervention that can be sustained at RLC following the completion of the funding period. Consistent with principles of community-engaged research, the investigators will share results with the Community Advisory Board (CAB), who will aid in interpretation and dissemination of results.

ELIGIBILITY:
Inclusion Criteria:

* female
* aged 18-74 years
* self-identifying as Black and/or Latina
* no personal history of breast cancer
* English- or Spanish-speaking
* having received a mammogram with normal results in the last 12 months
* ≥20% lifetime breast cancer risk per the NCI Breast Cancer Risk Assessment Tool (BCRAT)

Exclusion Criteria:

* aged <18 or ≥75
* pregnancy

Ages: 18 Years to 74 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Informed decisions about breast MRI | 1 month
  According to the Multidimensional Measure of Informed Choice, an informed decision is made with adequate knowledge and consistent with the respondent's preferences. Thus, two groups are classified as having made an informed decision: (1) those with adequate MRI knowledge, whose preferences align with screening with mammogram + MRI, and who intend to undergo MRI; and (2) those with adequate MRI knowledge, whose preferences align with screening with mammogram only, and who do not intend to undergo MRI. The knowledge, preferences, and intentions scores collected at T1 will be used to identify informed decisions.

SECONDARY OUTCOMES:
Decision Satisfaction | 1 month
  The Satisfaction With Decision (SWD) scale includes 6 items rated from "strongly disagree" (1) to "strongly agree" (5). Items are averaged to create a total score ranging from 1-5 (higher=greater satisfaction). Instructions will specify decisions about breast cancer screening.
Decisional Conflict | 1 month
  The low-literacy version of the Decisional Conflict Scale (DCS) includes 10 items rated as "yes" (0), "unsure" (2), or "no" (4). Items are summed and transformed to create total scores ranging from 0-100 (higher=more conflict). Instructions will specify decisions about breast cancer screening.

OTHER OUTCOMES:
MRI Knowledge | 1 month
  This breast MRI knowledge scale includes 10 true/false items based on the content of the breast MRI decision aid. Items are scored as correct (1) or incorrect (0); item scores are summed to create total scores (higher=greater knowledge). Adequate knowledge is specified as ≥50% correct.
Screening Preferences | 1 month
  Respondents will rate factors that are viewed as important by people deciding about breast cancer screening (e.g., length of procedure, false positives, cost, etc.) on a 12-point scale ranging from "not at all important" (0) to "extremely important" (11). Items are averaged to create are averaged to create a total score ranging from 0-11 (lower=preference for screening with mammogram only, higher=preference for screening with mammogram + breast MRI).
Screening Intentions | 1 month
  Participants will indicate screening intentions on a single item with a 7-point scale ranging from "mammogram only" (-3) to "mammogram + breast MRI" (3), with "unsure" as the mid-point (0).
Enacted Decision | 6 months
  Receipt of MRI (yes/no) will be assessed via EMR review.
Dosage/Fidelity | 1 month
  Self-reported receipt and use of the decision aid.
Preparation for Decision Making | 1 month
  The 10-item Preparation for Decision Making (PDM) Scale assesses opinions about the effect of the decision aid. Items are rated from "not at all" (1) to "a great deal" (5). Items are summed and transformed to create total scores ranging from 0-100 (higher=more prepared for decision making).
Decision Aid Bias | 1 month
  Participants will indicate whether the decision aid suggested that they should screen with mammogram (-1), screen with mammogram + breast MRI (1), or neither (0).

CONTACTS AND LOCATIONS:
Overall Officials: Claire C. Conley, PhD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes